CLINICAL TRIAL: NCT04686461
Title: Effect of Thymoquinone Extracted From Nigella Sativa in the Treatment of Arsenical Keratosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Farhana Nargis, MD, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2020/1642
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Keratotic Nodular Size

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nigella sativa seeds extract containing ointment intervention (Experimental): Nigella sativa seeds extract containing ointment dose- twice daily for 12 weeks
  Interventions: Drug: Nigella sativa seeds extract containing ointment intervention

INTERVENTIONS:
Drug: Nigella sativa seeds extract containing ointment intervention — Nigella sativa seeds extract containing ointment Nigella sativa seed extract, bee wax, white petrolatum, stearyl alcohol

SUMMARY:
Prepare an ointment from Nigella sativa seeds extract and apply it over palmer arsenical keratosis patient for 12 weeks. After than the effect of the ointment will be observed by measuring the keratotic nodular size before and after the intervention.

DETAILED DESCRIPTION:
Arsenicosis is a massive public health problem affecting thousands of people worldwide, especially India, West Bengal, and Bangladesh. In our country groundwater of estimated 59 administrative districts have been contaminated with high concentration of arsenic. Through this contaminated drinking water a large number of populations are chronically exposed to high concentration of arsenic. Arsenicosis is characterized by diffuse melanosis followed by hyperpigmentation and keratosis. Keratosis causes reduce working capacity that affects socioeconomic condition of the patient. Invasive skin lesions like squamous cell carcinoma, Bowen's disease, and basal cell carcinoma also caused by it. Keratosis can treated by several topical preparation like propylene glycol, salicylic acid, alpha-lipoic acid, neem leaf extract, solanum melongena extract, Azadirachta indica and oral preparation like zinc, antioxidant, and folic acid. This treatment procedure required longer time to relieve symptom and reduce patient's compliance. Nigella sativa is a well-known spice of Southeast Asia, especially in Bangladesh. It contains a yellow volatile oil, a fixed oil, protein, amino acid, reducing sugars, alkaloids, and minerals like potassium, sodium, phosphorus, and iron while zinc, magnesium, calcium, copper, and manganese are found in low level. Thymoquinone is a main pharmacologically active constituent of volatile oil of N. sativa. Other constituents of the volatile oil are thymol, thymohydroquinone, and dithymoquinone. These biologically active compounds possess antimicrobial, anti-inflammatory, antioxidant, immunological, antimetastatic, anti-diabetic activity. Study with Nigella sativa in the treatment of arsenical keratosis was done and found effective. Therefore, the study will be done to identification of compound that is isolated from Nigella sativa and its effect on moderate to severe arsenical keratosis. . After obtaining clearance from IRB, on the basis of selection criteria, 34 patients of arsenical keratosis will be enlisted from Bhanga Upazilla of Faridpur district, an arsenic affected area. The study will be an experimental study and conducted in Bangabandhu Sheikh Mujib Medical University. Nigella sativa extract will be collected by using n-hexane as a solvent and rotary evaporator. Thin Layer Chromatography (TLC), Nuclear Magnetic Resonance (NMR) and Infrared (IR) spectrometry of the extract will be done to identify compound. Cytotoxicity test of the extract will be analyzed by using brine shrimp bioassay. . Then a topical ointment will be prepared from Nigella sativa extract and supplied to the arsenical keratosis patient at two weeks interval. Instruction about the application of the ointment on keratotic lesion will be given to the patients. Adherence and side effects of the ointment will be monitored at regular interval over phone calls and during field visit. Keratotic nodular size will be measured before start and after completion of treatment. Photograph will also take before and after treatment. Improvement of the lesion will be measured by mean scoring of nodule and perception of patients about their improvement by using Likert Scale. Statistical analysis and results will be presented in tabulated forms and in different diagrams.

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 - 65 years
* Arsenical keratosis: Presence of moderate to severe keratosis (>5 mm) in both palms or soles
* Drinking arsenic-contaminated water (>50 µg/ L) for at least more than six months
* Patient did not receive topical application of any drug for the last three months
* Patient agreed to participate voluntarily
* Patient who understood the instruction of applying drug and could apply drug as per an instruction

Exclusion Criteria:

* Age <19 and >65 years
* Pregnant and nursing mother
* Patient who received any treatment of arsenicosis within the last three months
* Patient with skin diseases like atopic dermatitis, eczema, and psoriasis
* Any systemic disease, inflammatory disease and infectious condition that affected the skin, for example, diabetes mellitus, rheumatoid arthritis, systemic lupus erythematosus and hepatitis
* Food allergy to Nigella sativa

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Keratotic nodular size | 12 weeks
  Lesion size will be measured by slide calipers

CONTACTS AND LOCATIONS:
Overall Officials: Bangladesh Bhanga, Faridpur, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bhanga, Farīdpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No